CLINICAL TRIAL: NCT05226793
Title: Medication Use Evaluation for Enoxaparin in Hospitalized COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 054.PHA.2021.R
Record Dates: First submitted 2022-02-03; First posted 2022-02-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Retrospective chart review to be conducted at Methodist Richardson Medical Center (MRMC) in Richardson, TX. All adult patients hospitalized with COVID-19 on enoxaparin for DVT prophylaxis will be included. Collected data will be analyzed to determine the safety and effectiveness of the varying enoxaparin doses, and results will be presented at the American Society of Health-System Pharmacists Midyear conference in December 2022.

DETAILED DESCRIPTION:
Retrospective chart review to be conducted at Methodist Richardson Medical Center (MRMC) in Richardson, TX. All adult patients hospitalized with COVID-19 on enoxaparin for DVT prophylaxis will be included. Collected data will be analyzed to determine the safety and effectiveness of the varying enoxaparin doses, and results will be presented at the American Society of Health-System Pharmacists Midyear conference in December 2022.

EPIC will be queried for data for this medication use evaluation, including the patient's age, sex, weight/BMI, ICU status, maximum D-dimer level, enoxaparin dose received, development of DVT or PE, incidence and type of bleeding events, readmission status, and mortality. Other patient specific factors such as the CCI score, Padua score, and IMPROVE score will be calculated using online risk assessment tools.

To calculate the CCI score, a search function will be used to analyze the patient's health information in order to determine their age, history of myocardial infarction, congestive heart failure, peripheral vascular disease, stroke or transient ischemic attack, dementia, chronic obstructive pulmonary disease, connective tissue disease, peptic ulcer disease, liver disease, diabetes mellitus, kidney function, cancer status, blood dyscrasias, and HIV status to estimate their 10-year probability of survival.

To calculate the Padua score, each patient must be evaluated for cancer status, history of VTE, mobility status, history of thrombophilic conditions, recent trauma or surgery, age, heart and/or respiratory failure, acute myocardial infarction and/or respiratory failure status, acute infection and/or rheumatologic disorder, obesity, and ongoing hormonal treatment. If a patient scores a 4 or more, then pharmacologic prophylaxis would be indicated.

Lastly, to calculate each patient's bleeding risk, the IMPROVE bleeding risk assessment will be used. For this tool, the patient's age, gender, renal function, liver function, platelet count, ICU status, the presence of a central venous catheter, active gastrointestinal ulcer, history of bleeding in the previous three months, presence of rheumatic disease, and active malignancy are needed to calculate the risk. If the patient scores a 7 or higher on the assessment, they are at an increased risk for bleeding.

ELIGIBILITY:
Inclusion Criteria:

Effectiveness of intermediate-intensity vs standard prophylactic enoxaparin regimens on preventing DVT and/or PE in patients with COVID-19, measured using the following variables:

* Enoxaparin dose (appropriate for kidney function)
* Charlson comorbidity index (CCI) score
* Padua prediction score for risk of VTE
* IMPROVE [International Medical Prevention Registry on VTE] bleeding risk assessment score
* ICU status
* Number of thromboembolic events
* Length of stay
* Readmissions for DVT and/or PE
* In-hospital mortality with associated DVT or PE

Exclusion Criteria:

* Safety of intermediate-intensity vs standard prophylactic enoxaparin regimens in patients with COVID-19, measured using the following variables:

  * Bleeding events
  * Type of bleeding event

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients age 18 years or older hospitalized with COVID-19 on prophylactic/non-therapeutic enoxaparin from January 1, 2021 to January 31, 2021
  Patients that do not have any other indication for use of enoxaparin (i.e., active DVT/PE, atrial fibrillation, etc.)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Enoxaparin dose (appropriate for kidney function) | 2021-2022
  Enoxaparin dose
Charlson comorbidity index (CCI) score | 2021-2022
  (CCI) score
Padua prediction score for risk of VTE | 2021-2022
  Padua prediction score
IMPROVE [International Medical Prevention Registry on VTE] bleeding risk assessment score | 2021-2022
  IMPROVE [International Medical Prevention Registry on VTE] bleeding risk assessment score
ICU status | 2021-2022
  ICU status
Number of thromboembolic events | 2021-2022
  Number of thromboembolic events
Length of stay | 2021-2022
  Days
Readmissions for DVT and/or PE | 2021-2022
  Readmissions for DVT and/or PE
In-hospital mortality with associated DVT or PE | 2021-2022
  In-hospital mortality with associated DVT or PE

SECONDARY OUTCOMES:
Bleeding events | 2021-2022
  Bleeding events
Type of bleeding event | 2021-2022
  Type of bleeding event

CONTACTS AND LOCATIONS:
Overall Officials: Betina Daniel, PharmD, Principal Investigator — Methodist
Locations (1):
- Methodist Richardson Medical Center, Richardson, Texas, United States